CLINICAL TRIAL: NCT00185055
Title: The Relative Effects of Single Doses of Olmesartan Medoxomil, Irbesartan and Valsartan at High Dosage Levels on the Renin-Angiotensin-Aldosterone System in Healthy Normal Subjects
Brief Title: The Relative Effects of Olmesartan Medoxomil, Irbesartan and Valsartan on the Activity of the Blood Pressure Control System in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 866-448
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
Keywords: olmesartan; valsartan; irbesartan; renin-angiotensin-aldosterone system
MeSH Terms: interventions — Olmesartan Medoxomil; Irbesartan; Valsartan

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Irbesartan
Drug: Valsartan

SUMMARY:
To assess the effects of 3 blood pressure drugs, called angiotensin receptor blockers, on the blood pressure control systems in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 to 65
* In good health

Exclusion Criteria:

* Any serious health problems
* Positive test for HIV, Hepatitis B and C
* History of drug and alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-11; Study Completion 2005-02

PRIMARY OUTCOMES:
To characterize the plasma renin activity (PRA) and urinary aldosterone response patterns to single doses of olmesartan medoxomil, irbesartan, and valsartan compared to placebo in normal volunteers.